CLINICAL TRIAL: NCT01747434
Title: Complaints and Presumptive Diagnosis in a Danish Emergency Department
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Christian Backer Mogensen, Assistant Professor, University of Southern Denmark
Other Study IDs: SLB-ED-05-2012
Record Dates: First submitted 2012-12-07; First posted 2012-12-11 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Symptoms on Admission; Presumptive Diagnosis on Admission; Final Diagnosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Acute patients in Denmark are often admitted to Emergency Departments by their General Practitioner with a presumptive diagnosis.

The aim of this study is to evaluate the diagnostic value of the pre-admission presumptive diagnosis and to assess if the presumptive diagnosis could be replaced by a number of symptom-based groups.

ELIGIBILITY:
Inclusion Criteria:

* all acute patients admitted to emergency department

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all acute admissions to a Danish Emergency Department in 2010
Sampling Method: Probability Sample
Enrollment: 10070 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
action diagnosis | 0-48 hours after admission

CONTACTS AND LOCATIONS:
Locations (1):
- Kolding Hospital Emergency Department, Kolding, Denmark

REFERENCES:
- [Derived] Carter-Storch R, Olsen UF, Mogensen CB. Admissions to emergency department may be classified into specific complaint categories. Dan Med J. 2014 Mar;61(3):A4802. PMID 24814917